CLINICAL TRIAL: NCT05707637
Title: Bipolar Radio-frequency Ablation After Standard Unipolar Approach for Ventricular Arrhythmias Originating From the Base of the Heart. The BiUniVA Prospective Registry
Brief Title: Bipolar Radio-frequency Ablation After Standard Unipolar Approach - Prospective Registry.
Acronym: BiUniVA
Status: Recruiting | Type: Observational
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Prof. Piotr Kulakowski, Professor, Centre of Postgraduate Medical Education
Other Study IDs: 123/2022
Record Dates: First submitted 2023-01-08; First posted 2023-02-01 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Ventricular Arrythmia
Keywords: ventricular arrhythmia; unipolar ablation; bipolar ablation; base of the heart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VA group: Consecutive patients with VA originating from the base of the heart undergoing unipolar ablation
  Interventions: Other: Ablation

INTERVENTIONS:
Other: Ablation — Unipolar and bipolar ablation

SUMMARY:
Treatment of ventricular arrhythmias (VA) originating at the base of the heart may be challenging. Unipolar radio-frequency (RF) ablation is a standard approach to treat VA, however, it fails in 10 to 75% of patients, depending on the localization of VA. The main reason for unipolar ablation failure is the intramural location of the source of VA. In such patients, bipolar ablation may occur effective. However, there are no prospective studies or registries on consecutive patients wilt failed unipolar ablation, therefore, the proportion of candidates for bipolar ablation after failed unipolar approach is not known. Also, invasive electrophysiological parameters associated with successful unipolar and bipolar ablation have not been well established. It has been hypothesised that (1) bipolar ablation fails in 12-75% (mean 30%) of consecutive patients and these patients are candidates for bipolar ablation, (2) local ventricular signal precocity > 20 ms, unipolar signal without R wave and pace mapping 12/12 predict effective unipolar ablation but not bipolar ablation, (3) morphology of VA from surface ECG can identify patients with possible intramural localization, and (4) successful ablation results in improvement of quality of life (QoL).

Aims:

1. To assess how many patients after failed unipolar ablation need redo procedure with bipolar ablation (primary end-point)
2. To assess which intraprocedural electrophysiological parameters predict success during standard unipolar ablation (secondary endpoint)
3. To assess short term efficacy of bipolar ablation (secondary endpoint)
4. To assess one-month efficacy of bipolar ablation (secondary endpoint)
5. To assess which intraprocedural electrophysiological parameters predict success during redo bipolar ablation (secondary endpoint)
6. To evaluate the performance of ECG-based algorithms in predicting the localization / origin of VA, especially of transmural origin (secondary endpoint)
7. To assess the effects of ablation on QoL (secondary endpoint)Methods. The study group consists of all consecutive patients who underwent unipolar ablation of VA originating from the base of the heart in the Grochowski Hospital and collaborating centres. All these patients are referred to Grochowski Hospital for further follow-up and treatment if needed, including bipolar ablation if initial unipolar approach failed. In all patients acute and one-month efficacy of unipolar and bipolar ablation is assessed.

DETAILED DESCRIPTION:
Treatment of ventricular arrhythmias (VA) originating at the base of the heart may be challenging. Although such sites as right ventricular or left ventricular outflow tracts (RVOT and LVOT) or aortic cusps (AoCusps) are usually easy to access, other VA locations may be difficult to reach. They include arrhythmias originating close to the great cardiac vein (GCV), anterior interventricular vein (AIV) or those coming from above the pulmonary valve (PV). In addition, a significant proportion of these arrhythmias have their source of origin in the mid-myocardium and such sites are difficult to ablate from endocardium or epicardium using standard techniques. It has been estimated that the efficacy of standard unipolar radio-frequency (RF) ablation ranges from 80-90% in patients with typical RVOT arrhythmias to 75% in cases with VA originating from LVOT and as low as 25% in VA coming from the left ventricular (LV) summit.

Unipolar radio-frequency (RF) ablation is a standard approach to treat VA. When it fails, bipolar RF ablation may be an attractive alternative. Using this approach, RF energy travels between the tip of ablation electrode and the tip of another electrode, called return or passive electrode. By proper positioning of the electrodes in two adjacent structures, the site of VA origin may lay between the tips of these electrodes and high density RF current may effectively destroy the tissue responsible for VA. The most frequently used electrode locations for bipolar RF ablation are left pulmonic cusp (LPC), AoCusps, aorto-mitral continuity (AMC) and GCV.

It has been shown in animal model that bipolar ablation causes denser and larger lesions than standard unipolar approach. The lesions are also deeper, more transmural and created without steam pops as compared with unipolar RF ablation. Also, the perpendicular orientation of the electrodes tips as well as irrigated catheters rather than standard catheters are important for bipolar ablation safety and efficacy.

The bipolar approach is usually used when unipolar ablation fails. To date, only case reports and case series have been published showing improved outcome when bipolar ablation was used during redo procedures. However, no prospective registry was performed to establish how many patients with VA originating from the base of the heart require bipolar ablation and which invasive electrophysiological (EP) parameters predict failure of unipolar ablation and the need for bipolar approach. One ongoing registry does include consecutive patients and is heterogenous. In the current guidelines for VT ablation, the bipolar approach is only shortly mentioned as one of new and still experimental approaches. Also the performance of surface ECG criteria to predict intra-mural VA and effects of bipolar ablation of quality of life have not been established.

2. Hypothesis.

1. Unipolar ablation fails in a mean of 30% (12-75% depending on VA site), consecutive patients with VA originating from the base of the heart and these patients are candidates for bipolar ablation.
2. Local ventricular signal precocity > 20 ms, unipolar signal without R wave and pace mapping 12/12 predict effective unipolar ablation
3. Local signal precocity, unipolar signal and pace mapping do not predict efficacy of bipolar ablation,
4. Morphology of VA from surface ECG can identify patients with possible intramural localization of arrhythmia origin in whom initial unipolar ablation fails
5. Successful ablation results in improvement of quality of life (QoL) 3. Aim.

a. To assess how many patients after failed unipolar ablation need redo procedure with bipolar ablation (primary end-point) b. To assess which intraprocedural electrophysiological parameters predict success during standard unipolar ablation (secondary endpoint) c. To assess acute efficacy of bipolar ablation (secondary endpoint) d. To assess one-month efficacy of bipolar ablation (secondary endpoint) e. To assess which intraprocedural electrophysiological parameters predict success during redo bipolar ablation (secondary endpoint) f. To evaluate the performance of ECG-based algorithms in predicting the localization / origin of VA, especially of transmural origin (secondary endpoint) g. To assess the effects of ablation on QoL (secondary endpoint) Methods. Patients. The study group consists of all consecutive patients who underwent unipolar ablation of VA originating from the base of the heart in the Grochowski Hospital and collaborating centres. All these patients are referred to Grochowski Hospital for further follow-up and treatment if needed, including bipolar ablation if initial unipolar approach failed.

Electrophysiology study During EP study three EP parameters characterizing potential site for RF application are assessed. If surface ECG suggests right-sided focus - RVOT is firstly explored. If ECG suggests left-sided focus AoCusps, LVOT, GCV and possibly AIV are firstly explored. The EP parameters consist of (1) precocity of local V signal measured as a difference between the onset of the surface QRS complex (in lead with the earliest onset) and the onset of local bipolar V signal, and (2) presence or absence of R wave in the unipolar V signal. The third (3) parameter - pace-mapping, is also performed and expressed in the number of surface ECG leads with concordant pace-induced and spontaneous QRS morphology and also expressed in percentage of pace-matching in each lead, using dedicated software (EP Bard Lab System, US).

Unipolar ablation. Patients undergo ablation in light sedation using fentanyl and midazolam. In case of lack of PVC in patients with a history PVC only, isoproterenol infusion is used to facilitate PVC occurrence. In patients who undergo ablation due to VT, programmed ventricular stimulation is used to induce VT and in case of non-inducibility, isoproterenol infusion is used and programmed ventricular stimulation repeated to induce VT. In these patients stimulation is repeated at the end of procedure.

RF applications are performed at site with best EP parameters. If this ablation fails, no further attempts are made unless another site is almost as good as initial one and V signal exceeds surface QRS onset.

Ablation is considered acutely effective if no sVT is induced or >90% reduction of PVC or abolition of nsVT (in patients with nsVT) is achieved.

Ablation is considered acutely failed if all possible sites of VA are mapped: RVOT, PA, GCV, LVOT, AoCusp, AMC (mapping of AVI is not obligatory if placing of ablation electrode there is not feasible) and after RF applications VA is present or no applications were made (no place with good EP parameters were found).

All procedures are performed using Smarttouch Thermocool catheter, ablation index and electroanatomical Carto® 3 (Biosense Webster, Diamond Bar, CA, USA) 3D mapping system. The Smartablate or nGEN ablators are used. Energy settings are standard as usually used for various sites, ranging from 20 watts at AoCusps to 40 watts in LVOT. The power, temperature and duration of RF applications may differ between patients according to the clinical needs and circumstances.

Medium-term efficacy of unipolar ablation. Medium-term efficacy of unipolar ablations is based on 24-h Holter ECG performed 1 month after ablation without any antiarrhythmic drugs (beta blockers are allowed). Efficacy is defined as >90% reduction of PVC (from baseline Holter) and abolition of nsVT (in patients with nsVT before ablation). In patients with sVT - no sVT recurrence during one month.

Bipolar ablation. Bipolar ablation is performed in a patient with failed/unsuccessful initial unipolar ablation during with all accessible sites were mapped and EP parameters collected.

Bipolar ablation is performed using the Osypka and Carto 3 systems. The HAT500 (OSYPKA AG, Rheinfelden, Germany) generator enables to perform bipolar ablation using two ablation catheters. Power levels and impedance are recorded and displayed for both electrodes. Two open-irrigated 3.5mm or 4 mm tip mapping and ablation catheters are inserted in two adjacent locations. One ablation electrode is active and the second ablation catheter is passive (also named as return) catheter and is not visible on the electro-anatomical system screen during RF energy application.

In general, three sites for bipolar system can be used: (1) LPC, (2) GCV with its extension - AIV and (3) LVOT/AoCusps/AMC/MA. The sites for ablation electrodes positioning are chosen based on intracardiac signals (where local signals exceeds the most the onset of the QRS complex), presumed localization of intramural substrate (anatomical approach - focus should be located between the tips of active and return electrode) and safety issues (no coronary artery between the tips of electrodes based on repeated coronary angiography). Thus, the possible configurations include (1) LPC → LVOT/AoCusps/AMC/MA, (2) GCV → LVOT/AoCusps/AMC/MA or (3) LPC → GCV.

Optimal energy settings for bipolar ablation have not been yet established and are adjusted to the actual needs for effective and safe RF applications in a given patient.

Medium-term efficacy of bipolar ablation. Acute and long-term efficacy are the same as for unipolar ablation.

Coronary artery angiography. Coronary artery angiography is performed routinely during bipolar ablation and in selected patients undergoing unipolar approach (as needed). The radial or femoral artery access is used to enable repetitive contrast injections into the coronary vessels.

Assessment of quality of life. In addition, all patients will be asked to fill-in quality of life (QoL) questionnaires - before and 1 month after ablation. Two types of questionnaire will be used: the EuroQoL (EQ-5D) and the EHRA questionnaire which was developed for patients with atrial fibrillation, however, in this study it will used for patients with VA.

ELIGIBILITY:
Inclusion Criteria:

1. Baseline Holter ECG before initial unipolar ablation within 6 months prior to the procedure, performed without antiarrhythmic drugs (beta-blockers allowed).
2. Initial unipolar ablation of VA originating from the base of the heart (R in II, III and aVF) performed according to the standard scheme which includes detailed measurements of EP parameters at each examined and/or ablated site and inspection of all three regions (RVOT with PA, GCV and LVOT/AoCusps/AMC/MA) in cases with unsatisfactory EP parameters or failed ablation at first or second site.
3. Typical indications for ablation: a. > 10 000 PVC in 24-hour Holter ECG or b. > 10% PVC in 24-hour Holter ECG or c. less frequent but symptomatic PVC or d. at least 3 episodes symptomatic non-sustained ventricular tachycardia (nsVT) (>3 QRS evolutions) in Holter ECG, regardless of the amount of PVC or e. sustained ventricular tachycardia (sVT), regardless of nsVT or PVC
4. Written informed consent

Exclusion Criteria:

1. History of > 1 unipolar ablation for VA originating at the base of the heart
2. Lack of properly acquired EP parameters during baseline unipolar ablation
3. Lack of baseline Holter ECG performed < 6 months prior to initial unipolar ablation
4. Absence of typical indication for ablation
5. Lack of written informed consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with ventricular arrhythmias originating from the base of the heart undergoing first standard unipolar ablation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Candidates for redo bipolar ablation | 2 years
  The number and percentage of patients after failed unipolar ablation who need redo procedure with bipolar ablation

SECONDARY OUTCOMES:
Precosity of signal predicting unipolar ablation success | 2 years
  Local ventricular signal precocity in miliseconds
Unipolar recording predicting unipolar ablation success | 2 years
  Presence (yes or now) of unipolar recording without R wave
Pace-mapping predicting success of unipolar ablation | 2 years
  Number of leads with >95% pace-mapping
Acute efficacy of bipolar ablation | 2 years
  Number of PVC per minute at the end of bipolar ablation
Mid-term efficacy of bipolar ablation | 2 years
  Number and percentage of PVC during 24 hour ECG monitoring
Precosity of signal predicting bipolar ablation success | 2 years
  Local ventricular signal precocity in miliseconds
Unipolar recording predicting bipolar ablation success | 2 years
  Presence (yes or now) of unipolar recording without R wave
Pace-mapping predicting success of bipolar ablation | 2 years
  Number of leads with >95% pace-mapping
ECG criteria to predict origin of ventricular arrhythmia | 2 years
  Sensitivity (%) and specificity (%) of examined ECG criteria in predicting site of arrhythmia origin
Effects of ablation on QoL | 2 years
  Number of points in the EuroQoL (EQ-5D) and the EHRA questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kulakowski, MD PhD, Principal Investigator — Centre for Medical Postgraduate Education; Agnieszka Sikorska, MD PhD, Study Chair — Centre for Medical Postgraduate Education
Locations (1):
- Department of Cardiology, Postgraduate Medical School, Grochowski Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
On reasonable request, individual participant data will be availabe
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from 2023 to 2026
Access Criteria: individual request from a researcher

REFERENCES:
- [Result] Stec S, Sikorska A, Zaborska B, Krynski T, Szymot J, Kulakowski P. Benign symptomatic premature ventricular complexes: short- and long-term efficacy of antiarrhythmic drugs and radiofrequency ablation. Kardiol Pol. 2012;70(4):351-8. PMID 22528707
- [Result] Yamada T, Yoshida N, Doppalapudi H, Litovsky SH, McElderry HT, Kay GN. Efficacy of an Anatomical Approach in Radiofrequency Catheter Ablation of Idiopathic Ventricular Arrhythmias Originating From the Left Ventricular Outflow Tract. Circ Arrhythm Electrophysiol. 2017 May;10(5):e004959. doi: 10.1161/CIRCEP.116.004959. PMID 28500177
- [Result] Neira V, Santangeli P, Futyma P, Sapp J, Valderrabano M, Garcia F, Enriquez A. Ablation strategies for intramural ventricular arrhythmias. Heart Rhythm. 2020 Jul;17(7):1176-1184. doi: 10.1016/j.hrthm.2020.02.010. Epub 2020 Feb 20. PMID 32087355
- [Result] Koruth JS, Dukkipati S, Miller MA, Neuzil P, d'Avila A, Reddy VY. Bipolar irrigated radiofrequency ablation: a therapeutic option for refractory intramural atrial and ventricular tachycardia circuits. Heart Rhythm. 2012 Dec;9(12):1932-41. doi: 10.1016/j.hrthm.2012.08.001. Epub 2012 Aug 2. PMID 22863684
- [Result] Sauer PJ, Kunkel MJ, Nguyen DT, Davies A, Lane C, Tzou WS. Successful ablation of ventricular tachycardia arising from a midmyocardial septal outflow tract site utilizing a simplified bipolar ablation setup. HeartRhythm Case Rep. 2018 Nov 20;5(2):105-108. doi: 10.1016/j.hrcr.2018.11.002. eCollection 2019 Feb. No abstract available. PMID 30820408
- [Result] Futyma P, Santangeli P, Purerfellner H, Pothineni NV, Gluszczyk R, Ciapala K, Moroka K, Martinek M, Futyma M, Marchlinski FE, Kulakowski P. Anatomic approach with bipolar ablation between the left pulmonic cusp and left ventricular outflow tract for left ventricular summit arrhythmias. Heart Rhythm. 2020 Sep;17(9):1519-1527. doi: 10.1016/j.hrthm.2020.04.029. Epub 2020 Apr 26. PMID 32348845
- [Result] Futyma P, Sander J, Ciapala K, Gluszczyk R, Wysokinska A, Futyma M, Kulakowski P. Bipolar radiofrequency ablation delivered from coronary veins and adjacent endocardium for treatment of refractory left ventricular summit arrhythmias. J Interv Card Electrophysiol. 2020 Sep;58(3):307-313. doi: 10.1007/s10840-019-00609-9. Epub 2019 Aug 11. PMID 31402415
- [Result] Della Bella P, Peretto G, Paglino G, Bisceglia C, Radinovic A, Sala S, Baratto F, Limite LR, Cireddu M, Marzi A, D'Angelo G, Vergara P, Gulletta S, Mazzone P, Frontera A. Bipolar radiofrequency ablation for ventricular tachycardias originating from the interventricular septum: Safety and efficacy in a pilot cohort study. Heart Rhythm. 2020 Dec;17(12):2111-2118. doi: 10.1016/j.hrthm.2020.06.025. Epub 2020 Jun 26. PMID 32599177
- [Result] Igarashi M, Nogami A, Fukamizu S, Sekiguchi Y, Nitta J, Sakamoto N, Sakamoto Y, Kurosaki K, Takahashi Y, Kimata A, Komatsu Y, Machino T, Kuroki K, Yamasaki H, Aonuma K, Ieda M. Acute and long-term results of bipolar radiofrequency catheter ablation of refractory ventricular arrhythmias of deep intramural origin. Heart Rhythm. 2020 Sep;17(9):1500-1507. doi: 10.1016/j.hrthm.2020.04.028. Epub 2020 Apr 28. PMID 32353585
- [Result] Kany S, Alken FA, Schleberger R, Baran J, Luik A, Haas A, Ene E, Deneke T, Dinshaw L, Rillig A, Metzner A, Reissmann B, Makimoto H, Reents T, Popa MA, Deisenhofer I, Piotrowski R, Kulakowski P, Kirchhof P, Scherschel K, Meyer C. Bipolar ablation of therapy-refractory ventricular arrhythmias: application of a dedicated approach. Europace. 2022 Jul 15;24(6):959-969. doi: 10.1093/europace/euab304. PMID 34922350
- [Result] Cronin EM, Bogun FM, Maury P, Peichl P, Chen M, Namboodiri N, Aguinaga L, Leite LR, Al-Khatib SM, Anter E, Berruezo A, Callans DJ, Chung MK, Cuculich P, d'Avila A, Deal BJ, Della Bella P, Deneke T, Dickfeld TM, Hadid C, Haqqani HM, Kay GN, Latchamsetty R, Marchlinski F, Miller JM, Nogami A, Patel AR, Pathak RK, Saenz Morales LC, Santangeli P, Sapp JL Jr, Sarkozy A, Soejima K, Stevenson WG, Tedrow UB, Tzou WS, Varma N, Zeppenfeld K. 2019 HRS/EHRA/APHRS/LAHRS expert consensus statement on catheter ablation of ventricular arrhythmias: Executive summary. J Interv Card Electrophysiol. 2020 Oct;59(1):81-133. doi: 10.1007/s10840-019-00664-2. PMID 31960344